CLINICAL TRIAL: NCT05770141
Title: Laser Hemorrhoidoplasty Procedure Versus Open Surgical Hemorrhoidectomy
Brief Title: Laser Hemorrhoidoplasty Versus Open Surgical Hemorrhoidectomy in Second and Third Degree Piles
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ebram Nasser Hakim Boules, Doctor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: laser hemorrhoidoplasty
Record Dates: First submitted 2023-01-22; First posted 2023-03-15 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Hemorrhoids
MeSH Terms: conditions — Hemorrhoids

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LHP GROUP (Other): patients received Laser Hemorrhoidoplasty procedure
  Interventions: Procedure: laser hemorrhoidoplasty
- MM GROUP (Other): patients received conventional open surgical hemorrhoidectomy
  Interventions: Procedure: open surgical hemorrhoidectomy

INTERVENTIONS:
Procedure: laser hemorrhoidoplasty — A skin incision of 3 mm was made about 1 to 1.5 cm of distance from the anal verge at the base of each hemorrhoidal node. The probe was driven through the incision in the submucosal tissue until reaching the area underneath the distal rectal mucosa. Then, ten to twelve effective pulses (adjusted to respective node dimensions) were fired. Half of them were fired in the submucosal tissue, the others in the intra-nodal compartment determining the shrinkage of the hemorrhoidal piles. The anal wounds were left open. At the end of the procedure an anal tampon was positioned.
  Arms: LHP GROUP
Procedure: open surgical hemorrhoidectomy — The anodermal wedge was incised, eventually removing external fibrosis and/or skin tags when present. Upward dissection started at this level with en-bloc excision of mucosal and submucosal layers from the underlying internal anal sphincter up to the anorectal ring. A compressive haemostatic sponge was left in place for 12-24 hours.
  Arms: MM GROUP

SUMMARY:
The study aims to compare the pain , duration of intervention and long term outcomes of laser hemorrhoidoplasty versus open surgical hemorrhoidectomy

DETAILED DESCRIPTION:
Hemorrhoidal disease is ranked first among diseases of the rectum and large intestine, and the estimated worldwide prevalence ranges from 2.9% to 27.9%, of which more than 4% are symptomatic .

Age distribution demonstrates a Gaussian distribution with a peak incidence between 45 and 65 years with subsequent decline after 65 years .Men are more frequently affected than women .

The anorectal vascular cushions along with the internal anal sphincter are essential in the maintenance of continence by providing soft tissue support and keeping the anal canal closed tightly. Hemorrhoids are considered to be due to the downward displacement of suspensory (Treitz) muscle .

There are many treatments of hemorrhoids varying from medications and band ligation to stapled hemorrhoidopexy, laser photocoagulation, sclerotherapy, Doppler-guided artery ligation, and finally surgery .

The indications for the surgical treatment include the presence of a significant external component, hypertrophied papillae, associated fissure, extensive thrombosis or recurrence of symptoms after repeated RBL. The technique employed may be open (Milligan-Morgan) or closed (Ferguson) .

Post hemorrhoidectomy pain is the commonest problem associated with the surgical techniques. The other early complications are urinary retention (20.1%), bleeding (secondary or reactionary) (2.4%-6%) and subcutaneous abscess (0.5%). The long-term complications include anal fissure (1% -2.6%), anal stenosis (1%), incontinence (0.4%), fistula (0.5%) and recurrence of hemorrhoids .

The study aims to compare the pain , duration time of intervention and long term outcomes of laser hemorrhoidoplasty versus open surgical hemorrhoidectomy

ELIGIBILITY:
Inclusion Criteria:

* II-III hemorrhoidal disease
* failure of conservative treatment

Exclusion Criteria:

* grade IV
* acutely thrombosed haemorrhoids
* patients affected by IBD involving rectum or anus
* patients previously surgically treated for hemorrhoidal disease and the inability to complete study protocol

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Pain evaluation | 30 postoperative days
  postoperative pain assessment with Visual Analogue Scale Score, The VAS consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be').
bleeding | 30 postoperative days
  The timing of bleeding after hemorrhoidectomy varies, and can be generally divided into immediate and delayed.5 Immediate bleeding occurs within 24 to 48 hours of a procedure and is likely related to loss of control of the vascular pedicle. Delayed bleeding is defined as bleeding reported up to 2 weeks postprocedure, and is more often related to infection or local trauma , patients often report frequent passing of small to moderate amounts of clot and bright red blood starting after bowel movement.

SECONDARY OUTCOMES:
Presence of recurrence | 6 months
  Patients were considered to have recurrent hemorrhoidal symptoms when any of the following were recorded: bleeding, itching, pain or discomfort affecting patient's perception of quality of life, which could either be associated or not to prolapse recurrence.

OTHER OUTCOMES:
anal stenosis | 6 months
  Patients who experience anal stenosis describe constipation, bleeding, pain, and incomplete evacuation.

IPD SHARING:
Plan to Share IPD: Undecided